CLINICAL TRIAL: NCT00432211
Title: A Double Blind, Placebo Controlled, Randomised Trial to Investigate the Efficacy of Juvista (Avotermin) in the Prevention or Improvement of Scar Appearance Following Scar Revision Surgery.
Brief Title: Juvista (Avotermin) in the Prevention or Improvement of Scar Appearance Following Scar Revision Surgery.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovo (Industry)
Responsible Party: Renovo Ltd, Renovo Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-319-1009
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Complete Scar Excision
  Interventions: Drug: Avotermin
- 2 (Placebo Comparator): Staged Excision of scar
  Interventions: Drug: Avotermin

INTERVENTIONS:
Drug: Avotermin — Complete Excision:- On Day 0,Following wound closure the two outer segments of the wound will receive either Juvista or placebo.100µl of vehicle containing 200ng of Juvista will be injected per linear centimetre into both margins of one segment of the wound,and 100µl of vehicle alone (placebo) will be injected per linear centimetre into the other segment of the wound. There will be a central area (at least 3cm) of untreated wound between the two segments.The treatments will be re-administered to each wound segment (A and B) 24 hours after the first administration.
  Staged Excision On Day 0, the two end segments of the scar will be excised.Following wound closure each subject will receive 100µl of vehicle containing 200ng of Juvista per linear centimetre intradermally into one wound, and 100µl of vehicle alone (placebo) per linear centimetre into the other wound.The trial treatments will be re-administered to each wound 24 hours after the first administration.

SUMMARY:
This study is being undertaken to investigate the efficacy and safety of Juvista (given as an intradermal injection of 200ng/100µl per linear centimetre of wound margin) in the prevention or improvement of scar appearance when administered intradermally to approximated wound margins following surgical scar revision.

In addition, this study will compare the scar revision techniques of complete excision (excision of the entire scar during one surgical procedure) and staged excision (excision of the outmost segments and central core separately).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-85 years who have provided written informed consent.
* A body mass index between 15 and 35 kg/m2 .
* Subjects with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol.
* Female subjects of child bearing potential who are using method(s) of contraception acceptable to the Investigator and agree to do so from at least the screening visit until one month after administration of the final study dose.
* Subjects with linear scars that, in the opinion of the Investigator, are suitable for revision by excision and direct closure. The area of scar to be revised must be at least 5cm in length and have at least two comparable areas.
* Subjects, who, in the opinion of the Investigator have stabilised, mature scars.

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have history or evidence of keloid scarring.
* Subjects with scars for revision that cross a joint or are in close proximity to an anatomical structure, which could lead to distortion of the resultant scar.
* Subjects with additional scars less than 3cm away from the area to be revised.
* Subjects with a history of a bleeding disorder.
* Subjects with diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerability or efficacy.
* Subjects who have had surgery in the area to be excised within one year of Day 0.
* Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Subjects who on direct questioning and / or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing.
* Subjects with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Subjects who are taking, or have taken, any investigational drugs including Juvista within 3 months prior to the screening visit.
* Subjects who are taking regular, continuous, oral corticosteroid therapy.
* Subjects who, in the opinion of the Investigator, have significant ongoing psychiatric disorders, which may interfere with the trial assessments / visits.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects who are or who become pregnant up to and including Day 0 or who are lactating.
* In the opinion of the Investigator, a subject who is not likely to complete the trial for whatever reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Investigator scar assessment | up to 7 month visit
Patient scar assessment | up to 7 month visit
Independent scar assessment | up to month 7

SECONDARY OUTCOMES:
Local tolerability | up to month 7
Adverse events | up to month 7

CONTACTS AND LOCATIONS:
Overall Officials: D A McGrouther, FRCS MD, Principal Investigator — University of Manchester
Locations (1):
- Renovo Clinical Trials Unit, Manchester, United Kingdom

REFERENCES:
- [Derived] So K, McGrouther DA, Bush JA, Durani P, Taylor L, Skotny G, Mason T, Metcalfe A, O'Kane S, Ferguson MWJ. Avotermin for scar improvement following scar revision surgery: a randomized, double-blind, within-patient, placebo-controlled, phase II clinical trial. Plast Reconstr Surg. 2011 Jul;128(1):163-172. doi: 10.1097/PRS.0b013e318217429b. PMID 21701333